CLINICAL TRIAL: NCT03329950
Title: A Phase 1 Study of CDX-1140 as Monotherapy or in Combination in Patients With Advanced Malignancies
Brief Title: A Study of CDX-1140 (CD40) as Monotherapy or in Combination in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX1140-01; KEYNOTE-A23 (Other: Merck)
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Breast Cancer; Gastric Cancer; Renal Cell Carcinoma; Ovarian Cancer; Cholangiocarcinoma; Bladder Urothelial Carcinoma; Pancreatic Adenocarcinoma; Colorectal Cancer; Esophageal Cancer; Hepatic Cancer; Head and Neck Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Other Solid Tumors; Diffuse Large B-cell Lymphoma (DLBCL); Mantle Cell Lymphoma; Indolent B-cell Lymphomas; Non-Hodgkin Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Waldenstrom's Disease; Marginal Zone Lymphoma; Mucosa Associated Lymphoid Tissue; Small Lymphocytic Leukemia
Keywords: CDX-1140; Solid Tumors; Liver Cancer; GI Cancer; Kidney Cancer; Celldex; Monoclonal; Antibody; CD40; CD-40; Flt3l; CDX-301; Lung Cancer; Bile duct cancer; TNBC; RCC; Non-Hodgkin Lymphoma; Follicular Lymphoma; Dendritic cell; Keynote A-23; pembrolizumab; Keytruda; Chemotherapy; Gemcitabine; Nab-paclitaxel; CD40L; CD40 Ligand; Pancreas cancer; Metastatic pancreas cancer; Unresectable pancreas cancer; Stage IV pancreas cancer; Squamous cell cancer lung; Non-squamous cell cancer lung; Metastatic lung cancer; Stage IV lung cancer; Squamous cell cancer of head and neck; Stage IV cancer of head and neck; Throat cancer; Oropharyngeal cancer; Laryngeal cancer; Oral cancer; FLT3 Ligand; fms-like tyrosine kinase 3 ligand; KEYTRUDA®
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Stomach Neoplasms; Carcinoma, Renal Cell; Ovarian Neoplasms; Cholangiocarcinoma; Colorectal Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Head and Neck Neoplasms; Fallopian Tube Neoplasms; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Gastrointestinal Neoplasms; Kidney Neoplasms; Lung Neoplasms; Bile Duct Neoplasms; Hyper-IgM Immunodeficiency Syndrome; Pancreatic Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms | interventions — pembrolizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CDX-1140 (Experimental): Part 1: Eligible patients will receive CDX-1140, based on cohort assigned, in 4 week cycles until progression, intolerance, or two years of treatment.
  Interventions: Drug: CDX-1140
- CDX-1140 and CDX-301 (Experimental): Part 2: Eligible patients will receive CDX-1140, based on cohort assigned, in 4 week cycles until progression, intolerance or two years of treatment. A fixed dose of CDX-301 is injected once a day for five days before cycles 1 and 2 of CDX-1140.
  Interventions: Drug: CDX-1140; Drug: CDX-301
- CDX-1140 and pembrolizumab (Experimental): Part 3: Eligible patients will receive CDX-1140, based on cohort assigned, in 3 week cycles until progression, or intolerance, or two years of treatment. A fixed dose of pembrolizumab will also be given in 3 week cycles.
  Interventions: Drug: CDX-1140; Drug: pembrolizumab
- CDX-1140 and chemotherapy (Experimental): Part 4: Eligible patients will receive CDX-1140, based on cohort assigned, in 4 week cycles until progression, or intolerance, or two years of treatment. Chemotherapy will also be given according to standard of care.
  Interventions: Drug: CDX-1140; Drug: Chemotherapy

INTERVENTIONS:
Drug: CDX-1140 — CDX-1140 will be administered every 4 weeks in Parts 1, 2 and 4, and every 3 weeks in Part 3.
Drug: CDX-301 — CDX-301 will be injected once a day for five days before Cycles 1 and 2.
  Arms: CDX-1140 and CDX-301
Drug: pembrolizumab — pembrolizumab will be administered every 3 weeks.
  Other Names: KEYTRUDA®
  Arms: CDX-1140 and pembrolizumab
Drug: Chemotherapy — Gemcitabine and Nab-paclitaxel will be administered on Day 1, Day 8 and Day 15 of each 4 week Cycle.
  Arms: CDX-1140 and chemotherapy

SUMMARY:
This is a study to determine the maximum tolerated dose (MTD) for CDX-1140 (CD40 antibody), either alone or in combination with CDX-301 (FLT3L), pembrolizumab, or chemotherapy and to further evaluate its tolerability and efficacy in expansion cohorts once the MTD is determined.

DETAILED DESCRIPTION:
This study will determine the MTD of CDX-1140 while also evaluating the safety, tolerability and efficacy of CDX-1140 alone (Part 1) or in combination with CDX-301 (Part 2), pembrolizumab (Part 3), or chemotherapy (Part 4) in patients with cancer.

Eligible patients that enroll to the dose-escalation portion of the study will be assigned to one of several dose levels of CDX-1140. The dose-escalation part of the study will test the safety profile of CDX-1140, alone or in combination with CDX-301, pembrolizumab or chemotherapy and determine which dose(s) of CDX-1140 will be studied in the expansion portions of the study.

All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

ELIGIBILITY:
Key Inclusion Criteria:

1. Recurrent, locally advanced or metastatic melanoma (including mucosal and/or ocular), bladder/urothelial, non-small cell lung cancer, pancreatic adenocarcinoma, breast, colorectal, gastric, esophageal, renal cell, hepatic, ovarian fallopian or primary peritoneal carcinoma, head and neck, and cholangiocarcinoma. Additional tumor types (except primary CNS tumors) may be enrolled after discussion with, and approval from, the medical monitor.
2. Must have received all standard of care therapies (approved or unapproved) as deemed appropriate by the treating physician. Patients who refuse standard therapy are excluded from the study.
3. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 3 months following last treatment
4. Willingness to undergo a pre-treatment and on-treatment biopsy, if required.

Additional Inclusion Criteria for Part 1:

1. Advanced diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma, or indolent B-cell lymphoma are also eligible.
2. Lymphoma patients must have received ≥ 1 prior systemic therapy

Additional Inclusion Criteria for Part 3:

1. Patients must have documented progression while receiving anti-PD-1 or anti-PD-L1 based regimens for FDA approved indications
2. Patients cannot have received more than one anti-PD-1 or anti-PD-L1 based regimen

Additional Inclusion Criteria for Part 4:

1. Patients must have metastatic pancreatic adenocarcinoma, and have not received previous treatment in a metastatic setting

Key Exclusion Criteria:

1. History of severe hypersensitivity reactions to other monoclonal antibodies.
2. Previous treatment with any anti-CD40 antibody or with FLT3L.
3. Inadequate washout period from prior therapy as defined in the Protocol.
4. Major surgery within 4 weeks prior to study treatment.
5. Use of immunosuppressive medications within 4 weeks or systemic corticosteroids within 2 weeks prior to study treatment.
6. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers. For all other cancers, the patient must be disease-free for at least 3 years to be allowed to enroll.
7. Active, untreated central nervous system metastases.
8. Active autoimmune disease or documented history of autoimmune disease.
9. History of (non-infectious) pneumonitis or has current pneumonitis.
10. Active infection requiring systemic therapy, known infection of HIV, Hepatitis B, or Hepatitis C.

Additional Exclusion Criteria for lymphoma patients in Part 1:

1. Prior allogenic stem cell transplantation
2. Patients who have received autologous stem cell transplant ≤ 12 weeks prior to the first dose of study drug.

There are additional criteria your study doctor will review with you to confirm your eligibility for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of CDX-1140 as assessed by CTCAE v5.0 | From first dose through 30 days after last dose
  The rates of drug-related adverse events will be summarized and maximum tolerated dose will be determined.

SECONDARY OUTCOMES:
Objective Response Rate | Every 8-12 weeks, starting with first dose until disease progression, assessed up to approximately 1-3 years.
  The percentage of patients who achieved a confirmed complete response or partial response by evaluation criteria in solid tumors for immune-based therapeutics (iRECIST; for solid tumor patients) and the lymphoma response to immunomodulatory therapy criteria (LYRIC; for lymphoma patients).
Clinical benefit rate | Every 8-12 weeks, starting with first dose until disease progression, assessed up to approximately 1-3 years
  The percentage of patients who achieve best response of confirmed CR or PR, or stable disease (SD) for at least four months
Duration of Response | First occurrence of a documented objective response to disease progression or death (up to approximately 1-3 years)
  The interval from which measurement criteria are first met for CR or PR until the first date that progressive disease is objectively documented
Progression-free survival | From first dose to the first occurrence of disease progression or death due to any cause (up to approximately 1-3 years)
  The time from start of study drug to time of progression or death, whichever occurs first
Overall survival | The time from start of study drug to death from any cause (up to approximately 1-3 years)
  The time from start of study drug to death
Immunogenicity evaluation | Prior to each dose of study treatment and at treatment discontinuation, up to approximately 1-3 years
  Serum samples will be obtained for assessment of human anti-CDX-1140 and anti-CDX-301 antibodies
Pharmacokinetic evaluation | Prior to each study treatment, multiple timepoints after each study treatment, and at treatment discontinuation up to approximately 1-3 years
  CDX-1140 and CDX-301 concentrations will be measured

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - HonorHealth Research Insititute, Scottsdale, Arizona
  - Northside Hospital, Inc., Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center Research LLC, Canton, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital (RIH) The Miriam Hospital (TMH), Providence, Rhode Island
  - Houston Methodist, Houston, Texas